CLINICAL TRIAL: NCT05021965
Title: The Effectiveness of At-home , In-office and Combined Dental Bleaching System ：A Randomized Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, vice dean of school and hospital of stomatology, Fujian Medical University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 20210715
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Tooth Bleaching

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1: have two weeks of at-home tooth bleaching (Experimental): Participants will receive two weeks of at-home tooth bleaching with 10% Carbamide peroxide(Opalescence PF 10%) for the maxillary anterior teeth.
  Interventions: Procedure: different combined of tooth bleaching procedure
- group 2 : have two sessions of in-office tooth bleaching (Experimental): Participants will receive two sessions（with a 1- week interval ） of in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%)for the maxillary anterior teeth.
  Interventions: Procedure: different combined of tooth bleaching procedure
- group 3 : one week of at-home and then have one session of in-office tooth bleaching (Experimental): Participants will receive one week of at-home tooth bleaching with 10% Carbamide peroxide(Opalescence PF 10%) and then receive one session of in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%)for the maxillary anterior teeth.
  Interventions: Procedure: different combined of tooth bleaching procedure
- group 4 : one week of in-office and then have one session of at-home tooth bleaching (Experimental): Participants will receive one session of in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%) and a week later receive one week of at-home tooth bleaching with 10% Carbamide peroxide(Opalescence PF 10%)for the maxillary anterior teeth.
  Interventions: Procedure: different combined of tooth bleaching procedure

INTERVENTIONS:
Procedure: different combined of tooth bleaching procedure — The participants will be randomly allocated into 4 groups and receive different kind of tooth bleaching protocol.

SUMMARY:
This randomized controlled clinical trial aimed to investigate the effectiveness of at-home , in-office and combined dental bleaching system.

DETAILED DESCRIPTION:
The participants with at least one maxillary tooth demonstrating shade A3 or darker will be recruited and randomly allocated into 4 groups according to the different tooth bleaching protocol：at-home bleaching for group 1,in-office bleaching for group 2 ,combined bleaching for group 3 and group 4.Participates in group 1 will receive two weeks of at-home tooth bleaching （Lasts 14 days and at least 8 hours every day ）with 10% Carbamide peroxide(Opalescence PF 10%) , group 2 will receive two sessions （with a 1- week interval ）of in-office tooth bleaching with 40% hydrogen peroxide (Opalescence Boost PF 40%)，group 3 will receive one week of at-home tooth bleaching （Lasts 7 days and at least 8 hours every day ）and then the eighth day receive one session of in-office tooth bleaching , group 4 receive one session of in-office bleaching and lasts 7 days at-home bleaching start on the eighth day . Colour parameters (CIE L*, a*, b*) will be measured with a spectrophotometer (Vita Easyshade Advance 4.0) at baseline (T1), after the first bleaching session (T2), after the second bleaching session (T3), 1 month after the completion of bleaching (T4). CIEDE2000 colour difference (△E00), the Whiteness Index for Dentistry (WID) and Tooth sensitivity (TS) will also be calculated. The data will be statistically analysed through repeated ANOVA and Tukey's test (α = 0.05).

ELIGIBILITY:
Inclusion Criteria:

* patients between 18 and 30 years of age, with fully erupted upper and lower incisors and canines without dental or periodontal disease or restorations, and with at least one maxillary tooth presenting color score A3 or darker, as measured with the Vita Classical guide (Vita Zahnfabrik, Bad Sa # ckingen, Germany) ordered by brightness

Exclusion Criteria:

* patients with systemic diseases or oral mucosal disorders, previous bleaching treatment, patients undergoing orthodontic treatment, pregnant or lactating women , people with known allergy to the product ingredients, smokers, and alcohol abusers, had severe internal tooth discoloration (e.g. tetracycline stains), had bruxism or any other pathology that could cause TS (such as gingival recession or dentin exposure).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Change in tooth colour | six weeks
  Colour parameters (CIE L*, a*, b*) will be measured with a spectrophotometer (Vita Easyshade Advance 4.0). The color alteration after each session will be given by the differences between the values obtained at the sessions and the baseline (∆E).

SECONDARY OUTCOMES:
Tooth sensitivity evaluation | two weeks
  Using the visual analogue scale (VAS) record the Tooth sensitivity (TS) throughout the entire treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, PhD, Principal Investigator — Fujian Medical University, China
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No